CLINICAL TRIAL: NCT02508922
Title: Vitamin D3 for Autism Spectrum Disorder: a Randomized, Double-blind, Placebo-controlled Trial.
Brief Title: Trial of Vitamin D3 Supplementation in Paediatric Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: The National Children's Hospital, Tallaght (Other)
Responsible Party: Principal Investigator, Conor Kerley, Dietitian and Nutrition Scientist, University of Dublin, Trinity College
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: NCHVitDASD
Record Dates: First submitted 2015-07-24; First posted 2015-07-27 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D3 (Experimental): 2000iu vitamin D will be taken daily for 20 weeks.
  Interventions: Dietary Supplement: Vitamin D3
- Placebo (Placebo Comparator): Matching placebo drops will be taken daily for 20 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — 2,000iu vitamin D drops will be taken daily for 20 weeks
  Other Names: cholecalciferol
  Arms: Vitamin D3
Dietary Supplement: Placebo — Matching placebo drops will be taken daily for 20 weeks
  Arms: Placebo

SUMMARY:
To build on a recent case study and open label trial, the investigators want to find out if vitamin D supplementation can influence behavioural and core symptoms of autism.

DETAILED DESCRIPTION:
The investigators will assess behavioural and core symptoms of autism before and after 20 weeks of vitamin D supplementation in a double-blind, placebo-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Positive autism diagnostic observation schedule
* Stable medication regimen
* Tolerate phlebotomy

Exclusion Criteria:

* Unstable or very severe autism
* Epilepsy
* Renal/liver/gastrointestinal disease

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2015-09; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in stereotypic behaviour from the aberrant behaviour checklist | Day 1 and day 140
  A subscale derived from the validated aberrant behaviour checklist

SECONDARY OUTCOMES:
Change from baseline in serum 25-hydroxyvitamin D levels | Day 1 and day 140
  Total vitamin D levels
Change from baseline in serum calcium levels, corrected for albumin | Day 1 and day 140
  Total serum calcium levels indicating calcium balance.
Change from baseline in aberrant behaviour checklist | Day 1 and day 140
  A validated scale for use in autism
Change from baseline in cytokines | Day 1 and day 140
  Serum will be analysed for specific cytokines
Change from baseline in autoimmune markers | Day 1 and day 140
  Serum will be analysed for specific autoimmune markers
Change from baseline in behaviour Assessment System for Children - Second Edition | Day 1 and day 140
  A validated scale for use in autism
Change from baseline in repetitive behavior Scale - Revised | Day 1 and day 140
  A validated scale for use in autism
Change from baseline in Social Responsiveness Scale | Day 1 and day 140
  A validated scale for use in autism
Change from baseline in Developmental Disabilities-Children's Global Assessment Scale | Day 1 and day 140
  A clinical global impression of autism
Change from baseline in Vitamin D and Sun Questionnaire | Day 1 and day 140
  A scale assessing behaviour related to vitamin D

CONTACTS AND LOCATIONS:
Locations (3):
- Ireland (3):
  - National Children's Hopsital, Dublin, Dublin
  - Linn Dara and BeechPark, Dublin
  - Trinity College Dublin, Dublin

REFERENCES:
- [Background] Cannell JJ. Autism and vitamin D. Med Hypotheses. 2008;70(4):750-9. doi: 10.1016/j.mehy.2007.08.016. Epub 2007 Oct 24. PMID 17920208
- [Background] Eyles DW. Vitamin D and autism: does skin colour modify risk? Acta Paediatr. 2010 May;99(5):645-647. doi: 10.1111/j.1651-2227.2010.01797.x. Epub 2010 Mar 8. No abstract available. PMID 20219042
- [Background] Becker KG. Autism, immune dysfunction and Vitamin D. Acta Psychiatr Scand. 2011 Jul;124(1):74; author reply 74-5. doi: 10.1111/j.1600-0447.2011.01688.x. Epub 2011 Mar 13. No abstract available. PMID 21395563
- [Background] Kocovska E, Fernell E, Billstedt E, Minnis H, Gillberg C. Vitamin D and autism: clinical review. Res Dev Disabil. 2012 Sep-Oct;33(5):1541-50. doi: 10.1016/j.ridd.2012.02.015. Epub 2012 Apr 21. PMID 22522213
- [Background] Mostafa GA, Al-Ayadhi LY. Reduced serum concentrations of 25-hydroxy vitamin D in children with autism: relation to autoimmunity. J Neuroinflammation. 2012 Aug 17;9:201. doi: 10.1186/1742-2094-9-201. PMID 22898564
- [Background] Cannell JJ. Autism, will vitamin D treat core symptoms? Med Hypotheses. 2013 Aug;81(2):195-8. doi: 10.1016/j.mehy.2013.05.004. Epub 2013 May 29. PMID 23725905
- [Background] Cannell JJ, Grant WB. What is the role of vitamin D in autism? Dermatoendocrinol. 2013 Jan 1;5(1):199-204. doi: 10.4161/derm.24356. PMID 24494055
- [Background] Patrick RP, Ames BN. Vitamin D hormone regulates serotonin synthesis. Part 1: relevance for autism. FASEB J. 2014 Jun;28(6):2398-413. doi: 10.1096/fj.13-246546. Epub 2014 Feb 20. PMID 24558199
- [Background] Jia F, Wang B, Shan L, Xu Z, Staal WG, Du L. Core symptoms of autism improved after vitamin D supplementation. Pediatrics. 2015 Jan;135(1):e196-8. doi: 10.1542/peds.2014-2121. Epub 2014 Dec 15. PMID 25511123
- [Background] Saad K, Abdel-Rahman AA, Elserogy YM, Al-Atram AA, Cannell JJ, Bjorklund G, Abdel-Reheim MK, Othman HA, El-Houfey AA, Abd El-Aziz NH, Abd El-Baseer KA, Ahmed AE, Ali AM. Vitamin D status in autism spectrum disorders and the efficacy of vitamin D supplementation in autistic children. Nutr Neurosci. 2016 Oct;19(8):346-351. doi: 10.1179/1476830515Y.0000000019. Epub 2015 Apr 15. PMID 25876214
- [Derived] Kerley CP, Power C, Gallagher L, Coghlan D. Lack of effect of vitamin D3 supplementation in autism: a 20-week, placebo-controlled RCT. Arch Dis Child. 2017 Nov;102(11):1030-1036. doi: 10.1136/archdischild-2017-312783. Epub 2017 Jun 16. PMID 28626020